CLINICAL TRIAL: NCT02308735
Title: Fatty Acid Ethyl Esters in Meconium of Infants of Diabetic Mothers: a Pilot Trial
Acronym: FAEE-IDM
Status: Terminated | Type: Observational
Why Stopped: Technology has advanced beyond the applicability of the study
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 3948
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Infants of Diabetic Mothers
Keywords: gestation; diabetes; ethanol
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Urine sample, meconium sample, placental cord blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Control: Pregnant women without either gestational or pre-gestational diabetes mellitus (and their offspring).
  Interventions: Other: N/A - No intervention
- A1 IDM: Pregnant women with abnormal glucose tolerance test but normal fasting serum glucose levels (and their offspring).
  Interventions: Other: N/A - No intervention
- A2 IDM: Pregnant women with abnormal glucose tolerance test and fasting hyperglycemia (and their offspring).
  Interventions: Other: N/A - No intervention
- PGDM - IDM: Pregnant women with diabetes mellitus diagnosed prior to current pregnancy (and their offspring).
  Interventions: Other: N/A - No intervention

INTERVENTIONS:
Other: N/A - No intervention

SUMMARY:
Gestational diabetes mellitus (GDM) affects as many as 14% of women in the United States. Furthermore, the number of pregnant women with pregestational diabetes mellitus (PGDM) is also increasing, mainly due to an increase in the diagnosis of non-insulin dependent diabetes mellitus. A recent study demonstrated that 1.3% of pregnancies are now complicated by PGDM and that PGDM now comprises 21% of the diabetes that complicate gestations, which represents a two fold increase since 1999. One notable side effect of diabetes is an elevation of endogenous ethanol production, which in turn may result in a rise in fetal production of fatty acid ethyl ester (FAEE). FAEE found in meconium have been utilized as a marker of prenatal ethanol exposure. Therefore, FAEE elevation could call into question maternal claims of abstinence from alcohol during pregnancy. This study seeks to determine if meconium FAEE levels in the newborns of abstinent women with various classifications of diabetes mellitus are increased when compared to non-diabetic, abstaining controls.

DETAILED DESCRIPTION:
Researchers will approach four groups of pregnant women at 24-26 weeks when they present for routine obstetrical out-patient appointments:

1. Those with PGDM
2. Those with White's Class A1 GDM
3. Those with White's Class A2 GDM
4. Non-diabetic controls

The medical records of these women will be examined to determine self-reporting of any alcohol or other drug usage while pregnant; women who report any illicit drug use (or ethanol use) while pregnant will not be eligible for this study. A routine urine drug screen will further confirm this finding. Women who have not reported alcohol use during their pregnancy will be questioned regarding medication usage while pregnant, as some medications do contain small amounts of ethanol. Women who are judged to have not consumed alcohol during their pregnancies (intentionally or incidentally) would then be included in the study.

Demographic information about the mother would also be collected (age, parity, length of pregnancy), as would the mother's most recent glycosylated hemoglobin level; additionally, a glycosylated hemoglobin level will be drawn on our presumptive controls (to allow for covert gestational diabetes mellitus). This lab draw would be added to the mother's routine lab studies and would not require an additional venipuncture.

A second urine drug screen will be performed on the mother upon her admission to the University of Oklahoma Health Sciences Center for the delivery of her baby. If both screens are negative and the baby does not meet any of the exclusion criteria, the baby will be enrolled in the study.

The initial meconium from each baby of the recruited mothers will be gathered. Approximately 1 g of meconium will be collected, frozen, and evaluated for fatty acid ethyl ester analysis at the United States Drug Testing Laboratories, Inc. We will also be sending a dried blood spot from the baby which will be collected at the time of the baby's scheduled newborn screen. This dried blood spot will be evaluated for phosphatidylethanol, an ethanol by-product.

ELIGIBILITY:
Inclusion Criteria: (understood to include only abstemious women)

1. . Pregnant women expected to deliver between 37 and 41 weeks gestation (controls), and their babies
2. . Pregnant women expected to deliver between 37 and 41 weeks gestation who have class A1 diabetes mellitus, and their babies
3. . Pregnant women expected to deliver between 37 and 41 weeks gestation who have class A2 diabetes mellitus, and their babies
4. . Pregnant women expected to deliver between 37 and 41 weeks gestation who were diagnosed with diabetes mellitus prior to their pregnancy, and their babies.

Exclusion Criteria:

1. . Mothers who self-reported any alcohol or any illicit drug use during their pregnancy (and their babies)
2. . Mothers who had a positive drug screen at any point during their pregnancy (and their babies)
3. . Babies whose mothers suffered a placental abruption during their pregnancy.
4. . Babies whose mothers had inadequate prenatal care (defined as <3 prenatal clinic visits prior to admission for delivery)
5. . Non-English-speaking mothers
6. . Babies who pass meconium in utero.
7. . Babies born with multiple congenital anomalies or abdominal wall defects.

Max Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 1. Teetotaling pregnant women either without a diagnosis of diabetes (controls) or with a diagnosis of diabetes mellitus (either gestational or pregestational).
  2. The liveborn infants resulting from the concurrent pregnancies of the women listed above.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2014-03; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas C Dannaway, MD, Principal Investigator — Dept of Pediatrics
Locations (1):
- Children's Hospital of Oklahoma, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Bentley-Lewis R, Levkoff S, Stuebe A, Seely EW. Gestational diabetes mellitus: postpartum opportunities for the diagnosis and prevention of type 2 diabetes mellitus. Nat Clin Pract Endocrinol Metab. 2008 Oct;4(10):552-8. doi: 10.1038/ncpendmet0965. Epub 2008 Sep 9. PMID 18779843
- [Background] Bell R, Bailey K, Cresswell T, Hawthorne G, Critchley J, Lewis-Barned N; Northern Diabetic Pregnancy Survey Steering Group. Trends in prevalence and outcomes of pregnancy in women with pre-existing type I and type II diabetes. BJOG. 2008 Mar;115(4):445-52. doi: 10.1111/j.1471-0528.2007.01644.x. PMID 18271881
- [Background] Lawrence JM, Contreras R, Chen W, Sacks DA. Trends in the prevalence of preexisting diabetes and gestational diabetes mellitus among a racially/ethnically diverse population of pregnant women, 1999-2005. Diabetes Care. 2008 May;31(5):899-904. doi: 10.2337/dc07-2345. Epub 2008 Jan 25. PMID 18223030
- [Background] Pichini S, Marchei E, Vagnarelli F, Tarani L, Raimondi F, Maffucci R, Sacher B, Bisceglia M, Rapisardi G, Elicio MR, Biban P, Zuccaro P, Pacifici R, Pierantozzi A, Morini L. Assessment of prenatal exposure to ethanol by meconium analysis: results of an Italian multicenter study. Alcohol Clin Exp Res. 2012 Mar;36(3):417-24. doi: 10.1111/j.1530-0277.2011.01647.x. Epub 2011 Dec 14. PMID 22168178
- [Background] Bearer CF, Jacobson JL, Jacobson SW, Barr D, Croxford J, Molteno CD, Viljoen DL, Marais AS, Chiodo LM, Cwik AS. Validation of a new biomarker of fetal exposure to alcohol. J Pediatr. 2003 Oct;143(4):463-9. doi: 10.1067/S0022-3476(03)00442-6. PMID 14571221
- [Background] Ostrea EM Jr, Hernandez JD, Bielawski DM, Kan JM, Leonardo GM, Abela MB, Church MW, Hannigan JH, Janisse JJ, Ager JW, Sokol RJ. Fatty acid ethyl esters in meconium: are they biomarkers of fetal alcohol exposure and effect? Alcohol Clin Exp Res. 2006 Jul;30(7):1152-9. doi: 10.1111/j.1530-0277.2006.00131.x. PMID 16792562
- [Background] Otasevic V, Lazovic V, Spalevic M, Marinkovic O. [Endogenous alcohol in patients with diabetes and in patients with severe liver disease]. Med Glas. 1972 Nov;26(11):391-4. No abstract available. Serbian. PMID 4669769
- [Background] Simic M, Ajdukovic N, Veselinovic I, Mitrovic M, Djurendic-Brenesel M. Endogenous ethanol production in patients with diabetes mellitus as a medicolegal problem. Forensic Sci Int. 2012 Mar 10;216(1-3):97-100. doi: 10.1016/j.forsciint.2011.09.003. Epub 2011 Sep 25. PMID 21945304
- [Background] Peterson J, Kirchner HL, Xue W, Minnes S, Singer LT, Bearer CF. Fatty acid ethyl esters in meconium are associated with poorer neurodevelopmental outcomes to two years of age. J Pediatr. 2008 Jun;152(6):788-92. doi: 10.1016/j.jpeds.2007.11.009. Epub 2008 Jan 10. PMID 18492517
- [Background] Gareri J, Lynn H, Handley M, Rao C, Koren G. Prevalence of fetal ethanol exposure in a regional population-based sample by meconium analysis of fatty acid ethyl esters. Ther Drug Monit. 2008 Apr;30(2):239-45. doi: 10.1097/FTD.0b013e318167cfe5. PMID 18367988
- [Background] Zelner I, Shor S, Lynn H, Roukema H, Lum L, Eisinga K, Koren G. Clinical use of meconium fatty acid ethyl esters for identifying children at risk for alcohol-related disabilities: the first reported case. J Popul Ther Clin Pharmacol. 2012;19(1):e26-31. Epub 2012 Jan 10. PMID 22247425
- [Background] Bakhireva LN, Leeman L, Savich RD, Cano S, Gutierrez H, Savage DD, Rayburn WF. The validity of phosphatidylethanol in dried blood spots of newborns for the identification of prenatal alcohol exposure. Alcohol Clin Exp Res. 2014 Apr;38(4):1078-85. doi: 10.1111/acer.12349. Epub 2014 Feb 11. PMID 24511895

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Pregnant women without either gestational or pre-gestational diabetes mellitus (and their offspring).
  N/A - No intervention
- A1 IDM: Pregnant women with abnormal glucose tolerance test but normal fasting serum glucose levels (and their offspring).
  N/A - No intervention
- A2 IDM: Pregnant women with abnormal glucose tolerance test and fasting hyperglycemia (and their offspring).
  N/A - No intervention
- PGDM - IDM: Pregnant women with diabetes mellitus diagnosed prior to current pregnancy (and their offspring).
  N/A - No intervention
Period: Overall Study
Arm/Group | Control | A1 IDM | A2 IDM | PGDM - IDM
Started | 2 | 0 | 0 | 2
Completed | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 2
Not completed — Physician Decision | 2 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Study ended due to lack of funding
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | A1 IDM | A2 IDM | PGDM - IDM | Total
Number analyzed (Participants) | 2 | 0 | 0 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Samples were never sent for analysis due to lack of funding for study.
  years | 31 (1) |  |  | 28.5 (4.5) | 29.8 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  |  | 2 | 4
  Male | 0 |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0 | 0
  Asian | 0 |  |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0 | 0
  Black or African American | 0 |  |  | 0 | 0
  White | 2 |  |  | 2 | 4
  More than one race | 0 |  |  | 0 | 0
  Unknown or Not Reported | 0 |  |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  |  | 2 | 0

OUTCOME MEASURES:

1. Primary Outcome: Meconium Fatty Acid Ethyl Ester Concentration
Description: A measure of ethanol metabolites in the meconium of an infant.
Time Frame: Three months
Population: This study enrolled four mother/infant dyads but never had results due to low enrollment number
Arm/Group | Control | A1 IDM | A2 IDM | PGDM - IDM
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Phosphatidylethanol Level
Description: A measure of phosphatidylethanol, an ethanol metabolite, in the cord blood of an infant.
Time Frame: Three months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through four months.
Arm/Group | Control | A1 IDM | A2 IDM | PGDM - IDM
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0 | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/0 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT02308735/Prot_SAP_000.pdf